CLINICAL TRIAL: NCT02521987
Title: Port Size and Post-Operative Pain Perception by Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Elizabeth Mueller, M.D., Associate Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 207726
Record Dates: First submitted 2015-07-24; First posted 2015-08-13 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 8mm Port (Active Comparator): Participates will be randomized to have an 8 mm assistant port used during their surgery. The participate will be asked to specify the point that represents their level of perceived pain intensity and mark it on the scale at four time points: baseline pain prior to the procedure in the pre-operatively holding area, 4 to 6 hours post operatively, on Post Operative Day 1 (POD1). The final pain assessment will be at the two weeks postoperative clinic visit.
  Interventions: Procedure: 8mm port
- 12mm Port (Experimental): Participates will be randomized to have an 12mm assistant port used during their surgery. The participate will be asked to specify the point that represents their level of perceived pain intensity and mark it on the scale at four time points: baseline pain prior to the procedure in the pre-operatively holding area, 4 to 6 hours post operatively, on Post Operative Day 1 (POD1). The final pain assessment will be at the two weeks postoperative clinic visit.
  Interventions: Procedure: 12mm port

INTERVENTIONS:
Procedure: 8mm port — Participate in this arm will have their procedure performed with an 8mm laparoscopic port.
  Arms: 8mm Port
Procedure: 12mm port — Participate in this arm will have their procedure performed with a 12mm laparoscopic port.
  Arms: 12mm Port

SUMMARY:
The purpose of this study is to determine if there is a difference in pain perception by participants when the assistant port size varies by 50% (8 mm to 12 mm).

DETAILED DESCRIPTION:
Minimally invasive approaches trade a single longer incision for 4-5 smaller incisions that allow abdominal access and abdominal insufflation through "ports". The increase in operative times is mostly due to the need to pass suture, needles, cameras and instruments through the abdominal ports. While, it is intuitive that smaller abdominal ports will result in less pain at the incision site, the port size is also limited by instrument size and the size of the needle. When ports are smaller, it can take a little more time for a needle or instrument to be passed into the port.

There is a paucity of research comparing different port sizes as they relate to participate pain and operative time especially in a randomized controlled trial setting. The investigators goal would be to determine if there is a difference in pain perception by patients when the assistant port size varies by 50% (8 mm to 12 mm).

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic surgery for pelvic organ prolapse.
* proficiency in English .

Exclusion Criteria:

* Not proficiency in English
* Previous participation/randomization in the study at a previous visit
* Pregnant women cannot participate
* History of abdominal wall pain
* Chronic pain patients

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Participants will be asked to specify the point that represents their level of perceived pain intensity and mark it on the VAS at four time points. | 2 weeks post-op visit
  Measured with Visual Analog Scale (VAS) for pain at 1) baseline pain prior to the procedure in the pre-operatively holding area, 2) 4-6 hours post-operatively in the post-anesthesia care unit (PACU), 3) on post-operative day 1(POD1) and 4) once two weeks post operatively.

SECONDARY OUTCOMES:
What is the physician's perception of operative difficulty throughout the case? Determination of physician struggle and frustration will be documented. | Day of surgery
  This will be measured by recording the time the first suture is placed when the physician asks for the mesh, to the time the incision is closed.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Mueller, MD, Principal Investigator — Loyola University Health System
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

REFERENCES:
- [Background] Nygaard I, Bradley C, Brandt D; Women's Health Initiative. Pelvic organ prolapse in older women: prevalence and risk factors. Obstet Gynecol. 2004 Sep;104(3):489-97. doi: 10.1097/01.AOG.0000136100.10818.d8. PMID 15339758
- [Background] Olsen AL, Smith VJ, Bergstrom JO, Colling JC, Clark AL. Epidemiology of surgically managed pelvic organ prolapse and urinary incontinence. Obstet Gynecol. 1997 Apr;89(4):501-6. doi: 10.1016/S0029-7844(97)00058-6. PMID 9083302
- [Background] Geller EJ, Siddiqui NY, Wu JM, Visco AG. Short-term outcomes of robotic sacrocolpopexy compared with abdominal sacrocolpopexy. Obstet Gynecol. 2008 Dec;112(6):1201-1206. doi: 10.1097/AOG.0b013e31818ce394. PMID 19037026
- [Background] McDermott CD, Hale DS. Abdominal, laparoscopic, and robotic surgery for pelvic organ prolapse. Obstet Gynecol Clin North Am. 2009 Sep;36(3):585-614. doi: 10.1016/j.ogc.2009.09.004. PMID 19932417